CLINICAL TRIAL: NCT05028907
Title: Evaluation of Lacrimal Punctal Changes by Anterior Segment Optical Coherence Tomography AS-OCT After Topical Combined Antibiotics and Steroids Treatment in Cases of Inflammatory Punctual Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Mahmoud, clinical researcher, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S20-159
Record Dates: First submitted 2021-08-30; First posted 2021-08-31 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Ophthalmopathy , Lacrimal System
MeSH Terms: conditions — Eye Diseases | interventions — Chloramphenicol; dexamethasone 21-phosphate; tetrahydrozoline; Hypromellose Derivatives; alpha-Tocopherol; Polyethylene Glycols; Hyaluronic Acid; Polyethylene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group one (cases with inflamatory punctal stenosis treated with steroids and antibiotics) (Experimental): patients with inflammatory punctal stenosis were treated by steroids and antibiotics and evaluated by anterior segment optical coherence tomography before and after treatment
  Interventions: Drug: 5 mg chloramphenicol, 1 mg dexamethasone sodium phosphate, 0.25 mg tetryzoline hydrochloride, 2 mg Hydroxypropyl Methyl Cellulose, 10 mg α-tocopherol acetate and 8 mg macrogol 400).
- control group (Placebo Comparator): patients with inflammatory punctal stenosis received only preservative free tear substitutes
  Interventions: Drug: sodium hyaluronate, polyethylene and propylene glycol based) three times daily for three months

INTERVENTIONS:
Drug: 5 mg chloramphenicol, 1 mg dexamethasone sodium phosphate, 0.25 mg tetryzoline hydrochloride, 2 mg Hydroxypropyl Methyl Cellulose, 10 mg α-tocopherol acetate and 8 mg macrogol 400). — The patients were advised to apply the drops 5 times daily for the first week, three times daily for the next two weeks and one time daily for another one week. The patients were examined before treatment, one week, one month and three months later.
  Arms: group one (cases with inflamatory punctal stenosis treated with steroids and antibiotics)
Drug: sodium hyaluronate, polyethylene and propylene glycol based) three times daily for three months — The patients were advised to apply the drops 5 times daily for the first week, three times daily for the next two weeks and one time daily for another one week. The patients were examined before treatment, one week, one month and three months later.
  Arms: control group

SUMMARY:
Punctal stenosis is an important etiological factor that should be considered when assessing patients with epiphora. Anatomically, acquired punctal stenosis is a condition in which the external opening of the lacrimal canaliculus is narrowed or occluded and also can be accompanied by canalicular ductal stenosis.1,2. Defining an anatomical clear cut-off value for punctal stenosis is difficult due to wide variations in patients' demographics. Clinically, punctal stenosis is defined as a punctum size restricting tear drainage in the absence of distal tear drainage abnormalities.2 Acquired punctal stenosis can be involutional, inflammatory, infectious or idiopathic.3,4 Inflammatory endogenous causes include chronic blepharitis, dry eye disease and ocular cicatricial pemphigoid.3 Exogenous noxious stimuli may be chemical such as topical or systemic medications, or physical as irradiation or mechanical. The harmful effect of topical medications such as antiglaucomatous drops, dexamesathone, mitomycin-C and the systemic medications such 5-Fluorouracil or paclitaxel may be related to the medication themselves, the preservatives as benzalkonium chloride in the commercial preparations, or duration of treatment with those medications.3,5-9 The basic ultra-structure response to those various noxious stimuli is early punctal occlusion by edema which is followed by conjunctival overgrowth, keratinization of punctal walls and cicatricial punctal stenosis.

Although spectral-domain OCT is still being widely used on the retina, its anterior segment module is considered a new modality for imaging of proximal lacrimal excretory passage and tears meniscus height (TMH).

Recent studies showed the ability of using AS-OCT to differentiate between various punctal causes of epiphora and improve the understanding of the lacrimal punctal structure in vivo.10-12 The aim of this work is to evaluate the role of AS-OCT in evaluation the punctal changes after treatment by antibiotics and steroids.

DETAILED DESCRIPTION:
Punctal stenosis is an important etiological factor that should be considered when assessing patients with epiphora. Anatomically, acquired punctal stenosis is a condition in which the external opening of the lacrimal canaliculus is narrowed or occluded and also can be accompanied by canalicular ductal stenosis.1,2. Defining an anatomical clear cut-off value for punctal stenosis is difficult due to wide variations in patients' demographics. Clinically, punctal stenosis is defined as a punctum size restricting tear drainage in the absence of distal tear drainage abnormalities.2 Acquired punctal stenosis can be involutional, inflammatory, infectious or idiopathic.3,4 Inflammatory endogenous causes include chronic blepharitis, dry eye disease and ocular cicatricial pemphigoid.3 Exogenous noxious stimuli may be chemical such as topical or systemic medications, or physical as irradiation or mechanical. The harmful effect of topical medications such as antiglaucomatous drops, dexamesathone, mitomycin-C and the systemic medications such 5-Fluorouracil or paclitaxel may be related to the medication themselves, the preservatives as benzalkonium chloride in the commercial preparations, or duration of treatment with those medications.3,5-9 The basic ultra-structure response to those various noxious stimuli is early punctal occlusion by edema which is followed by conjunctival overgrowth, keratinization of punctal walls and cicatricial punctal stenosis.

Although spectral-domain OCT is still being widely used on the retina, its anterior segment module is considered a new modality for imaging of proximal lacrimal excretory passage and tears meniscus height (TMH).

Recent studies showed the ability of using AS-OCT to differentiate between various punctal causes of epiphora and improve the understanding of the lacrimal punctal structure in vivo.10-12 The aim of this work is to evaluate the role of AS-OCT in evaluation the punctal changes after treatment by antibiotics and steroids.

ELIGIBILITY:
Inclusion Criteria:

* Patients included aged 21 years or more who developed acquired inflammatory punctal edema and were complaining of epiphora. Epiphora of the included groups was grade2 according to Kashkoli's classification and grade 1:5 according to Munk's classification.

Exclusion Criteria:

* Patients excluded who had history of previous ocular and lacrimal surgery, trauma, lower lid margin malposition or laxity, dry eye (for control group), glaucoma, corneal abnormalities (abrasions, keratitis), congenital punctal anomalies, nasolacrimal duct obstruction, mucocele, pyocele were excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
widening of the punctum | 3 months
  the widening in the punctum after treatment which could be identified by anterior sehment optical coherence tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: immediatly and no end time
Access Criteria: punctal stenosis